CLINICAL TRIAL: NCT01018979
Title: A Phase II, Open-Label, Multi-Center Study to Evaluate the Safety, Pharmacokinetics, and Hematopoietic Stem Cell Mobilization of TG-0054 in Patients With Multiple Myeloma, Non-Hodgkin Lymphoma or Hodgkin Disease
Brief Title: Safety and PK/PD of TG-0054 in Multiple Myeloma, Non-Hodgkin Lymphoma and Hodgkin Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GPCR Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TG-0054-02
Record Dates: First submitted 2009-11-24; First posted 2009-11-25 (Estimated); Results first posted 2015-01-15 (Estimated); Last update posted 2021-05-11 (Actual); Status verified 2021-04

CONDITIONS: Multiple Myeloma; Non-Hodgkin Lymphoma; Hodgkin Disease
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hodgkin Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TG-0054 (2.24 mg/kg) (Experimental): TG-0054: 2.24 mg/kg TG-0054 administrated via 15-min IV infusion(allow a maximum of six leukapheresis sessions)
  Interventions: Drug: TG-0054 (2.24 mg/kg)
- TG-0054 (3.14 mg/kg) (Experimental): TG-0054: 3.14 mg/kg TG-0054 administrated via 15-min IV infusion(allow a maximum of six leukapheresis sessions)
  Interventions: Drug: TG-0054 (3.14 mg/kg)

INTERVENTIONS:
Drug: TG-0054 (2.24 mg/kg) — TG-0054: 2.24 mg/kg TG-0054 administrated via 15-min IV infusion(allow a maximum of six leukapheresis sessions)
  Arms: TG-0054 (2.24 mg/kg)
Drug: TG-0054 (3.14 mg/kg) — TG-0054: 3.14 mg/kg TG-0054 administrated via 15-min IV infusion(allow a maximum of six leukapheresis sessions)
  Arms: TG-0054 (3.14 mg/kg)

SUMMARY:
A phase II study to evaluate the safety, pharmacokinetics, and hematopoietic stem cell mobilization of TG-0054 in patients with multiple myeloma, non-Hodgkin lymphoma or Hodgkin disease.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 18 to 70 years of age inclusive
* Patients with confirmed pathology diagnosis of MM, NHL or HD
* Potential candidate for autologous stem cell transplantation at Investigator's discretion
* ≦ 2 prior regimens of cytotoxic chemotherapy (rituximab, thalidomide, and bortezomib will not be considered as cytotoxic chemotherapy)
* > 4 weeks since last cycle of chemotherapy prior to the study drug administration
* Total dose of melphalan received ≦ 200 mg in the most recent chemotherapy treatment
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Recovered from all acute toxic effects of prior chemotherapy at Investigator's discretion
* White blood cell (WBC) count ≧ 3.0 x 109/L on screening laboratory assessments
* Absolute neutrophil count ≧ 1.5 x 109/L on screening laboratory assessments
* Platelet count ≧ 100 x 109/L on screening laboratory assessments
* Serum creatinine ≦ 2.2 mg/dL on screening laboratory assessments
* Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and total bilirubin < 2 x upper limit of normal (ULN) on screening laboratory assessments
* Negative for human immunodeficiency virus (HIV)
* Adequate cardiac and pulmonary function to undergo leukapheresis at Investigator's discretion
* For females, one of the following criteria must be fulfilled:

  1. At least one year post-menopausal, or
  2. Surgically sterile, or
  3. Willing to use a double-barrier method [intrauterine device (IUD) plus condom, spermicidal gel plus condom] of contraception throughout the study
* Males must be willing to use a reliable form of contraception (use of a condom or a partner fulfilling the above criteria) from study Day 1 until 28 days after the last dose of TG-0054
* Able to provide the signed informed consent

Exclusion Criteria:

* Received radiation therapy around the pelvic or spinal area within 6 months prior to the study drug administration
* >10% bone marrow involvement of lymphoma in NHL patients
* Failed previous stem cell collection [failed to collect 2 x 106 CD34+ cells/kg within 4 apheresis sessions after receiving granulocyte colony-stimulating factor (G-CSF)]
* Patients who have undergone previous stem cell transplantation procedure
* Received G-CSF within 2 weeks prior to the study drug administration
* History of other cancer within the past 5 years excluding MM, NHL, HD, basal cell or squamous cell carcinoma of the skin
* History of other hematologic disorders including bleeding or thromboembolic disease
* History of poor and uncontrollable cardiovascular or pulmonary disease such as myocardial infarction, cardiac arrhythmias, transient ischemic attack, stroke or Chronic Obstructive Pulmonary Disease (COPD) patients hospitalized more than two times a year due to underlying disease
* Diagnosis of sickle cell anemia or documented sickle cell trait
* Uncontrollable malignancy with MM, NHL or HD, or carcinomatous meningitis, at Investigator's discretion
* Any infection required antibiotic treatment or unexplained fever above 38 °C within 3 days prior to dosing
* Pregnant or breast-feeding
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study
* Received any other investigational drug within 1 month before entering the study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2010-02; Primary Completion 2011-10 (Actual); Study Completion 2011-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tzeon-Jye Chiou, MD, Principal Investigator — Taipei Veterans General Hospital, Taiwan; Tso-Fu Wang, MD, Principal Investigator — Buddist Tzu Chi General Hospital; Sheng-Fung Lin, MD, Principal Investigator — Kaohsiung Medical University; Chih-Cheng Chen, MD, Principal Investigator — Chang Gung Memorial Hospital, Chiayi; Po-Nan Wang, MD, Principal Investigator — Chang Gung Memorial Hospital; Jih-Luh Tang, MD, Principal Investigator — National Taiwan University Hospital
Locations (6):
- Taiwan (6):
  - Chang-Gung Memorial Hospital Chiayi, Chiayi City
  - Buddist Tzu Chi General Hospital, Hualien City
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Chang-Gung Memorial Hospital Linkou, Linkou District
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 20 subjects were randomized. Among these, 19 subjects met all eligibility criteria and received at least one dose of TG-0054.
Period: Overall Study
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Started | 7 | 13 (A total of 20 subjects were randomized.)
Received at Least One Dose | 7 | 12
Completed | 4 | 3
Not Completed | 3 | 10
Not completed — Peak CD34+ cell count in PB < 10 cell/uL | 3 | 9
Not completed — Not received at least one dose | 0 | 1

BASELINE CHARACTERISTICS:
Population: 19 subjects met all eligibility criteria and received at least one dose of TG-0054.
Groups:
- Total: Total of all reporting groups
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg) | Total
Number analyzed (Participants) | 7 | 12 | 19
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.3 (15.5) | 52.4 (9.3) | 50.5 (11.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 11
  Male | 3 | 5 | 8
Height [Mean (Standard Deviation); unit: centimeters] | 162.7 (10.1) | 158.7 (8.6) | 160.2 (9.1)
Weight [Mean (Standard Deviation); unit: kilogram] | 67.3 (23.1) | 60.6 (10.2) | 63.1 (15.9)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/ meter^2] | 25.1 (6.0) | 24.0 (3.0) | 24.4 (4.2)
Diagnosis [Number; unit: participants]
  Multiple myeloma | 3 | 4 | 7
  Non-Hodgkin lymphoma | 3 | 7 | 10
  Hodgkin disease | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients Who Achieved Mobilization Success of Hematopoietic Stem Cells in Patients With Multiple Myeloma (MM), Non-Hodgkin Lymphoma (NHL) or Hodgkin Disease (HD).
Description: Patients who met the target CD34+ cell collection of ≧2 x 106 cells/kg after two apheresis sessions were classified as achieving mobilization success.
Time Frame: 1 week
Population: In TG-0054 (2.24 mg/kg) group, A total of 4 patients (2 with MM, 1 with NHL, and 1 with HD) underwent apheresis procedure.
  In TG-0054 (3.14 mg/kg) group, A total of 3 patients (1 with MM and 2 with NHL) underwent apheresis procedure.
Measure: Number; unit: participants
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 4 | 3
participants
  MM | 1 | 1
  NHL | 1 | 0
  HD | 0 | 0

2. Secondary Outcome: Maximum Plasma Concentration (Cmax) of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: According to the protocol, blood samples for PK assessment of TG-0054 were obtained from 6 consenting patients in each arm on study Day 1 at pre-dose, end of infusion, and 1 hr, 3 hr, 6 hr, 9 hr, 12 hr, 24 hr and 36 hrs after infusion.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
ng/mL | 20971 (6995) | 29665 (18583)

3. Secondary Outcome: Fold Increase of Circulating CD34+ Cell Counts in Peripheral Blood.
Time Frame: Baseline, 3 hours and 6 hours after infusion
Measure: Mean (Standard Deviation); unit: fold
Groups:
- Multiple Myeloma (MM): 7 patients with MM were enrolled.
- Non-Hodgkin Lymphoma (NHL) + Hodgkin Disease (HD): 10 patients and 2 patients with NHL and HD were enrolled, respectively.
- All Patients: All patents = MM + NHL + HD
Arm/Group | Multiple Myeloma (MM) | Non-Hodgkin Lymphoma (NHL) + Hodgkin Disease (HD) | All Patients
Number analyzed (Participants) | 7 | 12 | 19
fold
  Fold increase (3 hours after infusion) | 7.0 (5.9) | 6.1 (6.1) | 6.4 (5.9)
  Fold increase (6 hours after infusion) | 7.8 (7.2) | 7.8 (10.4) | 7.8 (9.1)
  Fold increase (Maximum increase) | 9.3 (7.5) | 10.3 (8.9) | 10.0 (8.4)
Statistical Analysis 1: Comparison: Multiple Myeloma (MM); Analyze whether the mean fold increase from the baseline to the peak time change was significant or not; Test type: Superiority or Other; p = 0.023, t-test, 2 sided — P values less than 0.05 are considered statistically significant in this study
Statistical Analysis 2: Comparison: Non-Hodgkin Lymphoma (NHL) + Hodgkin Disease (HD); Analyze whether the mean fold increase from the baseline to the peak time change was significant or not; Test type: Superiority or Other; p = 0.038, t-test, 2 sided — P values less than 0.05 are considered statistically significant in this study

4. Secondary Outcome: Time at Which Maximum Plasma Concentration is Observed (Tmax) of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
hr | 0.25 (0) | 0.25 (0)

5. Secondary Outcome: Terminal Elimination Half-life (t1/2) of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
hr | 4.65 (0.4) | 4.28 (0.6)

6. Secondary Outcome: Terminal Elimination Rate Constant (λz) of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: 1/hr
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
1/hr | 0.15 (0.01) | 0.16 (0.02)

7. Secondary Outcome: The Area Under the Plasma Concentration Time Curve (AUC) From 0 Hours to Time t of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 43610 (7034) | 55814 (12153)

8. Secondary Outcome: The Area Under the Plasma Concentration Time Curve (AUC) From 0 Hours to Infinity of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
hr*ng/mL | 43713 (7039) | 55920 (12170)

9. Secondary Outcome: Clearance (CL) of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/ hr/kg
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
mL/ hr/kg | 52.5 (9.4) | 58.6 (13.0)

10. Secondary Outcome: Volume of Distribution at the Terminal State (Vz) of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
mL/kg | 351 (62) | 366 (112)

11. Secondary Outcome: Volume of Distribution at Steady State (Vss) of TG-0054 in 12 Consented Patients With MM, NHL or HD.
Description: Plasma concentrations of TG-0054 were determinate by validated LC-MS/MS method.
Time Frame: 36 hrs after infusion
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Number analyzed (Participants) | 6 | 6
mL/kg | 179 (64) | 193 (76)

12. Secondary Outcome: Circulating CD34+ Cell Counts in Peripheral Blood.
Time Frame: Baseline, 3 hours and 6 hours after infusion
Measure: Mean (Standard Deviation); unit: cells/μL
Arm/Group | Multiple Myeloma (MM) | Non-Hodgkin Lymphoma (NHL) + Hodgkin Disease (HD) | All Patients
Number analyzed (Participants) | 7 | 12 | 19
cells/μL
  PB CD34+ count (Baseline) | 1.0 (0.7) | 0.9 (0.5) | 1.0 (0.6)
  PB CD34+ count (3 hours after infusion) | 5.7 (4.0) | 4.0 (2.1) | 4.6 (2.9)
  PB CD34+ count (6 hours after infusion) | 6.3 (3.9) | 4.3 (2.7) | 5.1 (3.3)
  PB CD34+ count (Maximum increase) | 7.8 (4.4) | 5.2 (3.7) | 6.5 (4.1)

ADVERSE EVENTS:
Time Frame: The whole study period, from Visit 1 (screening, day -14) to Visit 9 (7 days after the last dose)
Description: There were 8 serious AEs (SAE) reported that were all unrelated to study drug. No AEs led to discontinuation of study drug treatment and there were no deaths reported in this study.
Arm/Group | TG-0054 (2.24 mg/kg) | TG-0054 (3.14 mg/kg)
Serious Adverse Events (participants affected / at risk) | 2/7 | 6/12
Other Adverse Events (participants affected / at risk) | 6/7 | 8/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | TG-0054 (2.24 mg/kg) (N=7) | TG-0054 (3.14 mg/kg) (N=12)
ADMISSION FOR PREPARATION OF PERIPHERAL BLOOD STEM CELL HARVEST (Surgical and medical procedures) | 0 | 3 — Post-treatment SAE. Definitely not related to study drug
AUTOLOGOUS STEM CELL TRANSPLANT (Surgical and medical procedures) | 0 | 1 — Post-treatment SAE. Definitely not related to study drug
HOSPITALIZATION FOR BONE MARROW TRANSPLANTATION (Surgical and medical procedures) | 1 | 0 — Post-treatment SAE. Definitely not related to study drug
AUTOLOGOUS HEMATOPOIETIC STEM CELL TRANSPLANTATION (Surgical and medical procedures) | 1 | 0 — Post-treatment SAE. Definitely not related to study drug
TREATMENT OF NON-HODGKIN LYMPHOMA (Surgical and medical procedures) | 0 | 1 — Post-treatment SAE. Definitely not related to study drug
PEIPHERAL BLOOD STEM CELL HARVEST (Surgical and medical procedures) | 0 | 1 — Post-treatment SAE. Definitely not related to study drug
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TG-0054 (2.24 mg/kg) (N=7) | TG-0054 (3.14 mg/kg) (N=12)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) — Post-treatment AE. Probably related to study drug.
ABNORMAL DATA OF INCREASE BILIRUBIN (Investigations) | 1 (1) | 0 (0) — Post-treatment AE. Probably not related to study drug.
CARDIAC DISORDERS-OTHER:QT PROLONG AT 24HR-36HR AFTER INFUSION (Investigations) | 0 (0) | 1 (1) — Post-treatment AE. Possible related to study drug.
CHEST TIGHTNESS (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) — Post-treatment AE. Probably not related to study drug.
CLONIC OF RIGHT KNEE (Nervous system disorders) | 1 (1) | 0 (0) — Post-treatment AE. Definitely not related to study drug.
DIARRHEA (Gastrointestinal disorders) | 1 (1) | 1 (1) — Post-treatment AE. 1 probably related and 1 definitely related.
DIZZINESS (Nervous system disorders) | 2 (2) | 1 (1) — Post-treatment AE. 2 definitely not related and 1 possible related.
DRY COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Post-treatment AE. Definitely not related.
ECCHYMOSIS OVER FEMORAL PUNCTURE SITE (General disorders) | 0 (0) | 1 (1) — Post-treatment AE. Definitely not related to study drug.
EMESIS (Gastrointestinal disorders) | 0 (0) | 1 (1) — Post-treatment AE. Definitely not related to study drug.
FEVER (General disorders) | 0 (0) | 1 (1) — Post-treatment AE. Possible related to study drug.
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (3) | 0 (0) — Post-treatment AE. All possible related to study drug.
HYPERTENSION (Vascular disorders) | 0 (0) | 1 (1) — Post-treatment AE. Definitely not related to study drug.
HYPOCALCEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) — Post-treatment AE. Definitely not related to study drug.
HYPOCALCIUM (Metabolism and nutrition disorders) | 1 (2) | 0 (0) — Post-treatment AE. Definitely not related to study drug.
HYPOKALEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (1) — Post-treatment AE. Probably not related to study drug.
HYPOTENSION (Vascular disorders) | 0 (0) | 1 (1) — Post-treatment AE. Definitely not related to study drug.
HYPOTENSION BP 82/51MMHG (Vascular disorders) | 1 (1) | 0 (0) — Post-treatment AE. Possible related to study drug.
HYPOVOLEMIC HYPOTENSION BP 78/56MMHG (Vascular disorders) | 1 (1) | 0 (0) — Post-treatment AE. Possible related to study drug.
INCREASE ALANINE AMINOTRANS-FERASE (Investigations) | 1 (1) | 0 (0) — Post-treatment AE. Probably not related to study drug.
INCREASE ALPHA-GANNA GLUTAMYL TRANSPEPTIDASE (Investigations) | 1 (1) | 0 (0) — Post-treatment AE. Probably not related to study drug.
ITCHY SKIN (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Post-treatment AE. Probably not related to study drug.
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 2 (3) | 2 (2) — Post-treatment Ae. 3 possible related and 2 probably related.
LOW BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Post-treatment AE. Probably related to study drug.
MILD ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) — Post-treatment AE. Probably related to study drug.
MILD DIARRHEA (Gastrointestinal disorders) | 1 (1) | 0 (0) — Post-treatment AE. Probably related to study drug.
MILD DIZZINESS (Nervous system disorders) | 1 (1) | 0 (0) — Post-treatment AE. Possible related to study drug.
MILD HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) — Post-treatment AE. Possible related to study drug.
NAUSEA (Gastrointestinal disorders) | 1 (1) | 0 (0) — Post-treatment AE. Probably related to study drug.
NUMBNESS OF FACE (Nervous system disorders) | 0 (0) | 1 (2) — Post-treatment AE. Definitely not related to study drug.
NUMBNESS OF FACE AND PALM (Nervous system disorders) | 1 (1) | 0 (0) — Post-treatment AE. Definitely not related to study drug.
NUMBNESS OF FACE HANDS AND LEGS (Nervous system disorders) | 1 (1) | 0 (0) — Post-treatment AE. Definitely not related to study drug.
NUMBNESS OF LEGS AND LIPS (Nervous system disorders) | 1 (1) | 0 (0) — Post-treatment AE. Definitely not related to study drug.
NUMBNESS OF LIPS (Nervous system disorders) | 1 (1) | 0 (0) — Post-treatment AE. Definitely not related to study drug.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI needs to inform sponsor and asks for permission before he/she discusses or publishes trial results after the trial is completed.